CLINICAL TRIAL: NCT07026162
Title: Series Study on the Application of G Protein-Biased Receptor Agonist Oliceridine in Gynecological Surgery (2)：Effects of Oliceridine Versus Sufentanil on Postoperative Nausea and Vomiting After Gynecological Laparoscopic Surgery
Brief Title: Oliceridine on Postoperative Nausea and Vomiting in Gynecological Laparoscopic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: YanYing Xiao (Other)
Responsible Party: Sponsor-Investigator, YanYing Xiao, Associate Professor of the Department of Anesthesiology, the Second Xiangya Hospital, Central south University, Second Xiangya Hospital of Central South University
Organization: Second Xiangya Hospital of Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LYEC2024-0425
Record Dates: First submitted 2025-05-27; First posted 2025-06-18 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Gynecologic Surgical Procedures; Postoperative Nausea and Vomiting (PONV); Laparoscopy
Keywords: Laparoscopy; Gynecologic Surgical Procedures; postoperative nausea and vomiting; Oliceridine
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oliceridine group (Experimental): Anesthesia and analgesia with Oliceridine
  Interventions: Drug: Oliceridine
- Sufentanil group (Other): Anesthesia and analgesia with sufentanil
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Oliceridine — For gynecological laparoscopic surgery, general anesthesia was induced with Oliceridine at a dose of 0.06 mg/kg (Yichang Renfu Pharmaceutical Co., Ltd., China). Intraoperative analgesia was administered with a total dose of Oliceridine ranging from 0.1 to 0.15 mg/kg. Postoperatively, Oliceridine was administered through a patient-controlled analgesia (PCA) system.
  Other Names: TRV130; olinvyk
  Arms: Oliceridine group
Drug: Sufentanil — For gynecological laparoscopic surgery, general anesthesia was induced with Sufentanil at a dose of 0.3 µg/kg (Yichang Renfu Pharmaceutical Co., Ltd., China). Intraoperative analgesia was provided with a total dose of Oliceridine ranging from 0.5 to 0.8 µg/kg. Postoperatively, Sufentanil was administered through a patient-controlled analgesia (PCA) system.
  Arms: Sufentanil group

SUMMARY:
The aim of this clinical trial is to evaluate the impact of the analgesic Oliceridine on postoperative nausea and vomiting (PONV) following gynecological laparoscopic surgery. It will also assess the safety profile of Oliceridine. The trial seeks to address the following key questions:

Can Oliceridine reduce the incidence of postoperative nausea and vomiting (PONV) in gynecological laparoscopic surgery? Does the incidence of PONV differ between patients receiving Oliceridine and those receiving the commonly used analgesic sufentanil in gynecological laparoscopic surgery? Are there any opioid-related adverse reactions in gynecological laparoscopic surgery patients using Oliceridine?

Participants will:

Receive Oliceridine or sufentanil for anesthesia induction, maintenance, and postoperative pain management.

Vital signs during surgery and the occurrence of postoperative nausea and vomiting will be recorded.

Be followed up for at least 48 hours.

DETAILED DESCRIPTION:
Study Design:

This randomized, double-blind, parallel-controlled trial compares oliceridine versus sufentanil for anesthesia/analgesia in gynecologic laparoscopy at Second Xiangya Hospital. The study features:

1. Randomization: Computer-generated 1:1 allocation via sealed envelopes
2. Blinding: Triple-blinding (participants, clinicians, outcome assessors) maintained through: Identical drug preparations (volume/appearance-matched);Separation between anesthesia nurses preparing drugs and clinical/research teams
3. Control: Active comparator (sufentanil) reflecting current standard practice.

Technical Methodology：

1. Anesthesia Protocol: Standardized induction with midazolam (0.05-0.10 mg/kg), study drug (sufentanil 0.3 μg/kg vs oliceridine 0.06 mg/kg), propofol (1.5-2.0 mg/kg), and cisatracurium (0.2-0.3 mg/kg). Maintenance via TIVA: propofol (4-10 mg/kg/h) + remifentanil (0.1-0.2 μg/kg/min). Pre-incision/closure boluses: Study drug dosed per group (sufentanil 0.1-0.2 μg/kg vs oliceridine 0.02-0.04 mg/kg).
2. Analgesia Management: PCA pump configuration: Sufentanil group: 2 μg/kg in 100 mL NS; Oliceridine group: 0.4 mg/kg in 100 mL NS; Fixed adjuncts: ondansetron 8 mg + dexamethasone 10 mg.Demand dose: 2 mL (lockout 10 min), max 10 mL/h.
3. Rescue Protocols: Analgesia: Sufentanil 5 μg or oliceridine 0.2 mg IV PRN; PONV: Ondansetron 4 mg + dexamethasone 5 mg; haloperidol 1 mg if refractory.

Quality Assurance Measures:

Anesthesia depth monitoring: BIS-guided propofol titration; Hemodynamic stability: Protocolized management of hypotension (defined as MAP <65 mmHg); Data validation: 10% random audit of time-stamped outcomes (PACU discharge, bowel recovery).

Pharmacokinetic Considerations:

Oliceridine dosing based on morphine equivalence (1mg ≈ 5mg morphine); Adjusted intraoperative dosing to account for context-sensitive half-time differences vs sufentanil.

Statistical Approach: Sample size:

Powered for PONV incidence difference (α=0.05, β=0.2); Analysis: ITT principle with sensitivity analysis for protocol deviations; Covariate adjustment: Stratification by Apfel risk factors (female sex, non-smoking, PONV history, opioid use).

ELIGIBILITY:
Inclusion criteria:

1. Elective gynecological laparoscopic surgery;
2. Age 18-65 years;
3. ASA physical status I-III;
4. Body mass index (BMI) 18-30 kg/m².

Exclusion criteria:

1. Severe dysfunction of major organs such as the heart, lungs, or brain;
2. History of allergy to opioid drugs, propofol, soybeans, or eggs;
3. Recent use of sedatives, analgesics, or monoamine oxidase inhibitors;
4. History of alcohol abuse;
5. Obstructive sleep apnea syndrome;
6. Difficult airway;
7. Psychiatric or neurological disorders; communication disorders;
8. Women who are lactating or pregnant.

Withdrawal criteria:

1. Subject requests withdrawal or withdraws voluntarily;
2. Change in surgical method requiring combined gastrointestinal surgery;
3. Occurrence of allergy to the investigational drug or life-threatening complications;
4. Reoperation within 48 hours postoperatively due to bleeding or other factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting(PONV) | From the time of awakening to 48 hours postoperatively . Specially, at the moment of awakening, at the time of leaving the PACU, postoperative 2 hours, 6 hours , 12 hours, 24 hours and 48 hours.
  PONV will be assessed within 48 hours postoperatively in the ward by a blinded investigator. Subjects are required to use the simplified PONV impact scale to report whether any PONV events occurred in the past 48 hours and to provide a rating. (Q1. Have you experienced vomiting or symptoms of vomiting? If yes, how many episodes in total? Under what circumstances did it occur? Was any medication administered for treatment? Q2. Have you experienced nausea? If yes, did the sensation of nausea affect your daily activities? Was any medication administered for treatment?) Mild PONV is defined as mild nausea or a single vomiting episode caused by water or physical activity. Moderate PONV includes two vomiting episodes or significant nausea needing rescue therapy. Severe PONV is more than two vomiting episodes or requiring multiple doses of rescue therapy. Absence of symptoms requiring treatment is considered complete remission.

SECONDARY OUTCOMES:
Incidence of postoperative vomiting (POV) postoperative 48 hours | From the time of awakening to 48 hours postoperatively. Specially, at the moment of awakening, at the time of leaving the PACU, postoperative 2 hours, 6 hours , 12 hours, 24 hours and 48 hours.
  Occurrence of postoperative vomiting postoperative 48 hours
Rescue antiemetic medications | From awakening to 48 hours postoperatively
  Record rescue antiemetic medication use within 48 hours postoperatively
Postoperative Visual Analog Scale (VAS) score | From the time of awakening to 48 hours postoperatively . Specially, at the moment of awakening, at the time of leaving the PACU, postoperative 2 hours, 6 hours , 12 hours, 24 hours and 48 hours.
  Resting visual analog scale (VAS) pain scores within 48 hours postoperatively, measured using a 10 cm movable ruler with a numerical scale of 0-10 on the reverse side. The left end ("0") indicates no pain, while the right end ("10") represents unbearable severe pain.
Ramsay sedation score | Postoperative 2 hours
  Ramsay sedation score at 2 hours postoperatively: a score of 1 indicates agitation, 3 or 4 indicates somnolence, and 5 or 6 indicates excessive sedation
Sleep quality score | At the night of the surgery day, Day 0
  Patient sleep quality will be assessed using a numerical rating scale based on an 11-point Likert scale, ranging from 0 to 10. A score of 0 indicates complete insomnia and extremely poor sleep quality, while a score of 10 represents excellent sleep quality. Severe insomnia is defined as a score of 0-3, moderate insomnia as 4-6, and good sleep quality as 7-10.
Quality of Recovery-15 (QOR-15) score | Preoperative, postoperative day 1, and postoperative day 3, respectively
  A score of 0 indicates extremely poor quality of recovery, while a score of 150 indicates excellent quality of recovery. Assessments will be conducted preoperatively, on postoperative day 1, and on postoperative day 3.
The time of the first postoperative bowel gas passage | From end of surgery until first postoperative passing of gas, assessed up to 72 hours.
  The time from the end of surgery to the first postoperative passing of gas
Time staying in the PACU | From PACU arrival until discharge, assessed up to 6 hours.
  The time from the patient's arrival to discharge from the PACU
Intraoperative hypotension | From anesthesia induction until PACU discharge, assessed up to 6 hours.
  Hypotension is defined as a mean arterial pressure (MAP) less than 65 mmHg lasting for one minute, during the surgery from the anesthesia induction until the patient leaves the PACU.

OTHER OUTCOMES:
Patient demographic characteristics | Baseline, preoperative
  Patient demographic characteristics including age, height, weight, BMI, ASA classification, smoking history, previous history of PONV, history of motion sickness, surgical history, history of hypertension, history of diabetes, among others.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD will be available when the last participant's follow-up is completed, and there is no time limit for its usage.
Access Criteria: Contact the author at any time.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT07026162/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT07026162/ICF_001.pdf